CLINICAL TRIAL: NCT02889107
Title: Long-term Use Benefits of Personal Frequency-modulated Systems for Speech in Noise Perception in Stroke Patients With Auditory Processing Deficits- 'a Non-randomised
Brief Title: Auditory Rehabilitation in Stroke Patients With Auditory Processing Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Responsible Party: Principal Investigator, Doris-Eva Bamiou, Reader & Consultant in Audiovestibular Medicine, University College, London
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 11/LO/1675
Record Dates: First submitted 2016-08-23; First posted 2016-09-05 (Estimated); Last update posted 2016-09-05 (Estimated); Status verified 2016-08

CONDITIONS: Auditory Processing Disorder, Central; Stroke
MeSH Terms: conditions — Language Development Disorders; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- standard care (No Intervention): Patients received standard listening strategies for 10 weeks
- intervention (Experimental): Patients received an assistive listening device (personal frequency modulated systems) for 10 weeks
  Interventions: Other: personal frequency modulated systems

INTERVENTIONS:
Other: personal frequency modulated systems — patients used personal frequency modulated systems for at least 4 hours daily for 10 weeks
  Other Names: FM systems
  Arms: intervention

SUMMARY:
This study aimed to evaluate long term benefits in speech reception in noise, after daily 10 week use of an assisting listening device (personal frequency-modulates systems) , in non-aphasic stroke patients with auditory processing deficits.

DETAILED DESCRIPTION:
Stroke can affect all levels of the auditory pathway. Approximately one in five stroke survivors report severe difficulties when listening to speech-in-noise, despite normal hearing, attributed to abnormal processing of sounds within the brain, and these individuals are more likely to experience communication difficulties in poor acoustic environments, The patient with significant auditory deficits and functional limitations may require a range of rehabilitation and remediation approaches. Several studies conclusively demonstrate substantial improvements in speech recognition in noise when using personal frequency-modulated (FM) systems. These devices are used to improve speech perception in noise in adults with neurological disorders including stroke with good immediate benefits. However, the long-term benefits of FM systems in stroke patients has not been studies. In this research study the investigators aimed to investigate the long term benefits in speech reception in noise in non-aphasic stroke patients and measure the potential improvement in unaided speech in background noise performance after 10 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Clinical history of ischaemic stroke verified by brain magnetic resonance imaging (MRI)
* Diagnosis of auditory processing disorders
* Normal pure-tone audiogram

Exclusion Criteria:

* Severe aphasia
* Significant psychiatric illnesses

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2013-04; Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
The signal-to-noise ratio (SNR) benefit for speech in noise (reported in decibel, dB) | week 1
  Patients are tested in a sound attenuated booth (the crescent of sound) with nine audio stands, an equipment cabinet, and a testing station for the assessment of spatial-listening skills. A 'Speech in noise' test was used. In this test, recorded spoken sentences are presented from straight ahead (0°) while noise is also coming from 90° to the left or right from the participant, who is asked to repeat the sentence. The number of keywords successfully repeated is recorded and repetition of at least three keywords per sentence is required to judge correct performance. The level of the sentences and the background noise are adaptively varied to estimate the signal-to-noise ratio (SNR) for 50% correct performance. The test was conducted with the participant using the frequency modulated systems (aided condition) or not using the frequency modulated systems (unaided condition). The level of SNR is reported in dB.

SECONDARY OUTCOMES:
The signal-to-noise ratio (SNR) benefit for speech in noise (reported in decibel, dB) | week 10
  Patients are tested in a sound attenuated booth (the crescent of sound) with nine audio stands, an equipment cabinet, and a testing station for the assessment of spatial-listening skills. A 'Speech in noise' test was used. In this test, recorded spoken sentences are presented from straight ahead (0°) while noise is also coming from 90° to the left or right from the participant, who is asked to repeat the sentence. The number of keywords successfully repeated is recorded and repetition of at least three keywords per sentence is required to judge correct performance. The level of the sentences and the background noise are adaptively varied to estimate the signal-to-noise ratio (SNR) for 50% correct performance. The test was conducted with the participant using the frequency modulated systems (aided condition) or not using the frequency modulated systems (unaided condition). The level of SNR is reported in dB.

CONTACTS AND LOCATIONS:
Overall Officials: Doris-Eva Bamiou, PhD, Principal Investigator — University College, London
Locations (1):
- University College London Hospitals, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Koohi N, Vickers D, Warren J, Werring D, Bamiou DE. Long-term use benefits of personal frequency-modulated systems for speech in noise perception in patients with stroke with auditory processing deficits: a non-randomised controlled trial study. BMJ Open. 2017 Apr 7;7(4):e013003. doi: 10.1136/bmjopen-2016-013003. PMID 28389484